CLINICAL TRIAL: NCT04028869
Title: Clinical Observation of Long-term Efficacy and Safety of Glycyrrhizic Acid Preparation in the Treatment of Autoimmune Liver Disease
Brief Title: Clinical Observation of Long-term Efficacy and Safety of Glycyrrhizic Acid Preparation in the Therapy of Autoimmune Liver Disease
Status: Completed | Type: Observational
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Director of the Second Division of Liver Diseases, Beijing Ditan Hospital
Other Study IDs: DTXY018
Record Dates: First submitted 2019-07-20; First posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Autoimmune Liver Disease
Keywords: Autoimmune liver disease; glycyrrhizic acid; liver function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Glycyrrhizin preparation treatment group: Clinical effect of glycyrrhizic acid preparation for 144 weeks of autoimmune liver disease and safety during treatment
  Interventions: Drug: Glycyrrhizic acid preparation

INTERVENTIONS:
Drug: Glycyrrhizic acid preparation — To analyze the clinical effect of glycyrrhizic acid preparation for autoimmune liver disease for 144 weeks and the safety during treatment

SUMMARY:
This study was a retrospective clinical observation cohort study. All patients with autoimmune liver disease treated with glycyrrhizic acid preparations in the Department of Liver Diseases, Department of Liver Diseases, Beijing Ditan Hospital, Capital Medical University, were enrolled. Clinical follow-up data including demographics, hematuria, and liver and kidney were collected. Functional, electrolyte blood glucose, PTA, erythrocyte sedimentation rate, serum AFP and other clinical biochemical indicators and autoantibodies, special proteins and liver imaging (liver ultrasound) examination. The clinical effect of glycyrrhizic acid preparation for the treatment of autoimmune liver disease for 144 weeks and the safety during treatment were analyzed.

DETAILED DESCRIPTION:
This study was a retrospective clinical observation cohort study. All patients with autoimmune liver disease treated with glycyrrhizic acid preparations in the Department of Liver Diseases, Department of Liver Diseases, Beijing Ditan Hospital, Capital Medical University, were enrolled. Clinical follow-up data including demographics, hematuria, and liver and kidney were collected. Functional, electrolyte blood glucose, PTA, erythrocyte sedimentation rate, serum AFP and other clinical biochemical indicators and autoantibodies, special proteins and liver imaging (liver ultrasound) examination. The clinical effect of glycyrrhizic acid preparation for the treatment of autoimmune liver disease for 144 weeks and the safety during treatment were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients with autoimmune liver disease: All enrolled autoimmune liver diseases meet the diagnostic criteria of China's Consensus on Diagnosis and Treatment of Autoimmune Liver Disease (2015);
* 2) no hormones and / or immunosuppressants and other liver protection drugs;
* 3) Sign the written informed consent form.

Exclusion Criteria:

* 1) Combine other hepatitis virus (HCV, HDV) infections;
* 2) viral liver disease;
* 3) HIV infection;
* 4) long-term alcohol abuse and / or other liver damage drugs;
* 5) mental illness;
* 6) Evidence of liver tumors (liver cancer or AFP > 100 ng/ml);
* 7) decompensated cirrhosis;
* 8) Serious diseases such as heart, brain, lung, kidney, etc. can not participate in long-term follow-up;
* 9) There are hormones and / or immunosuppressants and other liver protection drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with autoimmune liver disease: All enrolled autoimmune liver diseases meet the diagnostic criteria of China's Consensus on Diagnosis and Treatment of Autoimmune Liver Disease (2015);
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
The ratio of sustained biochemical responses | at 96 weeks and 144 weeks after treatment
  The ratio of sustained biochemical responses at 96 weeks and 144 weeks after treatment with glycyrrhizic acid preparation in patients with autoimmune liver disease

SECONDARY OUTCOMES:
The incidence of decompensated liver cirrhosis and liver cancer and its complications | at 96 and 144 weeks after treatment
  The incidence of decompensated liver cirrhosis and liver cancer and its complications at 96 and 144 weeks after treatment with glycyrrhizic acid in patients with autoimmune liver disease

CONTACTS AND LOCATIONS:
Overall Officials: Yao Xie, Doctor, Principal Investigator — liver disease center, Beijing Ditan Hospital
Locations (1):
- liver disease center, Beijing Ditan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No